CLINICAL TRIAL: NCT05154812
Title: Based on the Comprehensive Evaluation System of Platelet Count/Splenic Length-diameter Ratio to Explore the Efficacy of Yang Yin Fu Zheng Jie Du Therapy in Delaying the Progression of HBV Associated Hepatocellular Carcinoma
Brief Title: Yang Yin Fu Zheng Jie Du Therapy in HBV Associated Hepatocellular Carcinoma Based on the Platelet Count/Splenic Length-Diameter Ratio
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Zhiyun Yang, Archiater, Professor, Beijing Ditan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BJDH-YZY
Record Dates: First submitted 2021-12-08; First posted 2021-12-13 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-12

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yang Yin Fu Zheng Jie Du therapy (Experimental)
  Interventions: Drug: Yang Yin Fu Zheng Jie Du therapy
- Routine medical care (Placebo Comparator)
  Interventions: Drug: Routine medical care

INTERVENTIONS:
Drug: Yang Yin Fu Zheng Jie Du therapy — Yang Yin Fu Zheng Jie Du is a Chinese herbal compound.
  Arms: Yang Yin Fu Zheng Jie Du therapy
Drug: Routine medical care — Routine medical care
  Arms: Routine medical care

SUMMARY:
Clinical research of Yang Yin Fu Zheng Jie Du therapy in HBV associated Hepatocellular Carcinoma based on the platelet count/splenic length-diameter ratio.The purpose of this study is to establish the efficacy evaluation system combined with platelet/splenic length-diameter ratio, and to clarify the effect of this method on relieving hepatitis B cirrhosis and delaying the progression of Hepatocellular Carcinoma.

ELIGIBILITY:
Inclusion Criteria:

Meet the criteria of hepatocellular carcinoma Patients who tested positive for hepatitis B surface antigen (HBsAg) for >6 months Liver function grade child-Pugh A/B Patients who have agreed to select local treatment according to the Guidelines for the Diagnosis and Treatment of Primary Liver Cancer (2017) TCM syndrome differentiation belongs to deficiency of qi and Yin, stasis and toxin accumulation syndrom Informed consent from the patient.

Exclusion Criteria:

Patient with other hepatitis virus infections or alcoholic liver, autoimmunity liver, primary biliary cirrhosis, genetic metabolic liver disease, and previous liver transplantation; Serious problem of heart, lung, brain, blood and other important organs; Patients with metastatic liver cancer; Pregnant or child breast feeding women; Mental or cognitive disorders; Who are allergic to the study drug.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Tumor progression rate | 1 year

SECONDARY OUTCOMES:
Overall survival rate | 1 year
Progression-free survival rate | 1 year
Median time to tumor progression | 1 year
Complete response rate | 1 year
the platelet count/splenic length-diameter ratio | 1 year
quality of life (QOL) questionnaire | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Zhiyun Yang, doctor, Beijing, Beijing Municipality, China